CLINICAL TRIAL: NCT02949492
Title: Low Dose IL-2 to Expand Endogenous Regulatory T-cells and Achieve Tolerance in Liver Transplantation
Brief Title: Low-dose IL-2 for Treg Expansion and Tolerance (LITE)
Acronym: LITE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LITE-01
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2018-03

CONDITIONS: Transplantation; Liver Diseases
Keywords: Liver; Transplant; Immunosuppression
MeSH Terms: conditions — Liver Diseases | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IL-2 arm (Experimental): Liver recipients <50 years old and 2-6 years after transplantation will receive IL-2 and gradually discontinue their immunosuppressive medication
  Interventions: Drug: IL-2 (interleukin 2)

INTERVENTIONS:
Drug: IL-2 (interleukin 2) — Low-dose IL-2 will be initiated while study participants remain on a calcineurin inhibitor immunosuppressant. Following 4 weeks of treatment, participants showing at least a 2-fold increase in peripheral blood absolute Treg numbers, stable liver function and no adverse effects will undergo a liver biopsy to exclude sub-clinical graft damage, and subsequently will initiate immunosuppression withdrawal. Low-dose IL-2 will be maintained for a total of 6 months.
  Other Names: Proleukin

SUMMARY:
Regulatory T cells (Tregs) suppress cytopathic immune responses and inhibit transplant rejection. Our goal is to exploit the Treg suppressive properties to induce transplantation tolerance. In contrast to effector T cells, Tregs constitutively express the high affinity IL-2 receptor, which makes them exquisitely sensitive to very low-doses of IL-2. We propose here to conduct a phase IV clinical trial in which we will test the capacity of low-dose IL-2 to promote the selective expansion of endogenous Tregs in liver transplant recipients at the time immunosuppressive drugs are being discontinued. We expect this will promote Treg accumulation within the transplanted liver, shift the balance between effector T cells and Tregs, and facilitate the development of operational tolerance in patients unlikely to reach this state spontaneously. We expect the trial to start shortly after the initiation of the project and to provide robust evidence on the efficacy of IL-2 within 47 months.

DETAILED DESCRIPTION:
Transplantation remains the most successful treatment for end-stage organ failure, but the need to administer life-long immunosuppression (IS) to prevent rejection limits patient survival. Liver transplantation is the only transplantation setting in which a sizeable proportion of patients spontaneously develop "operational tolerance", a phenomenon defined by the maintenance of stable graft function in the absence of destructive immune responses without the need of IS. Unfortunately this phenomenon preferentially develops in elderly recipients and several years after transplantation. To maximize the benefit derived from IS discontinuation there is a need to find strategies to intentionally induce tolerance in young recipients in whom accumulated IS toxicity has not yet occurred. Our studies have revealed that successful IS discontinuation is associated with a transient intra-graft immune regulatory response with preferential accumulation of regulatory T cells (Tregs). This suggests that short-term enhancement of Treg numbers and/or function at the time of IS withdrawal may facilitate the acquisition of tolerance in patients who are not predisposed to spontaneously develop it. IL-2 is a cytokine that is essential for the optimal development, survival and function of Tregs. Several clinical studies have shown that low-dose IL-2 preferentially expands Tregs and is safe and efficacious in patients with autoimmunity or GVHD. In these studies, Treg frequency increased up to 2 to 8-fold without significant changes in the number of effector T cells. Our objective is to investigate if administration of a short-course of low dose IL-2 to liver transplant recipients facilitates the discontinuation of IS. We propose to conduct a phase II, safety and efficacy, prospective, single-arm clinical trial in which liver recipients <50 years old and 2-6 years after transplantation will receive IL-2 and gradually discontinue their IS medication.

ELIGIBILITY:
Inclusion Criteria:

1. Adult liver transplant recipients 2-6 years post-transplant and age <50 years;
2. Recipient of single organ transplant only;
3. Liver function tests: direct bilirubin and ALT <2 x ULN at the screening visit;
4. On calcineurin inhibitor (CNI) based IS; with or without one of the following: Low dose mycophenolic acid (≤ 1080 mg daily), mycophenolate mofetil (MMF ≤ 1500 mg daily), or azathioprine (≤ 150 mg daily);
5. Provision of written informed consent.

Exclusion Criteria:

1.1. Serum positivity for HCV-RNA at screening; 2. Serum positivity for HIV-1 infection, HBV surface antigen or HBV-DNA at screening; 3. Active liver or systemic immune-mediated disease in which IS discontinuation is inadvisable (autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cirrhosis); 4. Acute or chronic rejection within the 52 weeks prior to screening; 5. GFR <40 mL/min (to mitigate the risk of worsening renal failure should rejection occur and high level of CNI be required); 6. The need for chronic anti-coagulation that cannot be safely discontinued to safely perform for a liver biopsy; 7. Screening liver biopsy showing signs of clinically significant histological damage will preclude continuation in the trial; 8. Maintenance immunosuppressive therapy with a mTOR inhibitor (sirolimus or everolimus); 9. Active infection or malignancy; 10. Inability to comply with study directed treatment; 11. Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial (including severe cardiac disease, severe respiratory disease with O2 blood saturation <92%, any other major organ dysfunction, and Eastern Cooperative Oncology Group (ECOG) performance status of ECOG > 1).

12. Participation in another IMP study within 3 months from consent; 13. Any known allergy or intolerance to the IMP components; 14. Pregnancy or lactation; 15. Lack of effective methods of contraception for women and men of childbearing potential; 16. Hypersensitivity to Proleukin or to any of the excipients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Discontinuation of immunosuppression drugs | 12 months post IS withdrawal
  The primary objective is to determine the capacity of a short course of low-dose IL-2 to facilitate the complete discontinuation of immunosuppressive drugs in liver recipients 2-6 years after transplantation.

SECONDARY OUTCOMES:
Proportion of tolerant participants remaining free of rejection | 12 months post IS withdrawal
  Measures of rejection in patients (incidence, severity, timing, steroid resistant rejection, chronic rejection) and to investigate if liver transplant recipients under IS become operationally tolerant over time.
Development of serum anti-HLA antibodies | 12 months post IS withdrawal
  To determine if the presence of donor-specific anti-HLA antibodies influence the success of IS withdrawal, and whether IS withdrawal promotes the development of anti-HLA antibodies in liver transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, Principal Investigator — King's College London
Locations (1):
- Alberto Sanchez-Fueyo, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim TY, Perpinan E, Londono MC, Miquel R, Ruiz P, Kurt AS, Kodela E, Cross AR, Berlin C, Hester J, Issa F, Douiri A, Volmer FH, Taubert R, Williams E, Demetris AJ, Lesniak A, Bensimon G, Lozano JJ, Martinez-Llordella M, Tree T, Sanchez-Fueyo A. Low dose interleukin-2 selectively expands circulating regulatory T cells but fails to promote liver allograft tolerance in humans. J Hepatol. 2023 Jan;78(1):153-164. doi: 10.1016/j.jhep.2022.08.035. Epub 2022 Sep 7. PMID 36087863